CLINICAL TRIAL: NCT06521359
Title: Role of Follicular Helper and Follicular Regulatory T Cells in Hashimoto's Thyroiditis
Brief Title: Role of Follicular T Cells in Hashimoto's Thyroiditis
Status: Not yet recruiting | Type: Observational
Sponsor: Omnia Ahmed Nafea Mohamed (Other)
Responsible Party: Sponsor-Investigator, Omnia Ahmed Nafea Mohamed, doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: flow cytometry in Hashimoto
Record Dates: First submitted 2024-07-22; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Hashimoto's Thyroiditis
MeSH Terms: conditions — Hashimoto Disease | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case
  Interventions: Device: flow cytometry
- control
  Interventions: Device: flow cytometry

INTERVENTIONS:
Device: flow cytometry — Two ml of peripheral venous blood samples will be collected in heparinized tubes from patients and controls for assessment of levels of TFH and TFReg cells by flow cytometry.

SUMMARY:
Measure the frequency of Follicular helper Tcells and Follicular regulatory T cells in peripheral blood samples in Hashimoto's pts in comparison with control.

DETAILED DESCRIPTION:
Hashimoto thyroiditis, also known as chronic autoimmune thyroiditis and chronic lymphocytic thyroiditis, is an autoimmune disease in which thyroid cells are destroyed via cell and antibody-mediated immune processes. It is the most common cause of hypothyroidism in developed countries. In contrast, the most common cause of hypothyroidism worldwide is an inadequate dietary intake of iodine. The pathophysiology of Hashimoto thyroiditis involves the formation of antithyroid antibodies that attack the thyroid tissue, causing progressive fibrosis. The diagnosis can be challenging, and consequently, the condition is sometimes not diagnosed until late in the disease process. The most common laboratory findings demonstrate elevated thyroid-stimulating hormone (TSH) and low thyroxine (T4) levels, coupled with increased antithyroid peroxidase (anti-TPO) antibodies and antithyroglobulin (anti-Tg) antibodies .

Recent years have shown that Hashimoto thyroiditis development depends on an immune defect in an individual with genetic susceptibility together with environmental factors .

ELIGIBILITY:
Inclusion Criteria:

- The study will include 45 Hashimoto's patients attending the out clinics of Endocrinology Department of Assiut university hospital. In addition, 45 healthy blood donors will be included as controls. The diagnosis of hashimoto's thyroiditis will be determined according to the criteria of American Thyroid Association;

* Having symptoms of hypothyroidism, and a blood test shows an underactive thyroid gland [an elevated thyroid stimulating hormone (TSH) level with or without a low thyroid hormone (free T4 or total T4) level].
* have elevated thyroid antibody levels.
* ultrasound examination demonstrating characteristic heterogeneous echotexture.
* results of thyroid fine needle aspiration (FNA) examinations meeting HT cytology diagnostic criteria.

Exclusion Criteria:

* -We should exclude other causes of thyroiditis, such as De Quervain's thyroiditis, Riedel's thyroiditis, and suppurative thyroiditis and also exclude other autoimmune diseases for example; type1 diabetes&Rheumatoid arthritis,and other diseases which cause hypothyroidism as carcinoma and surgery.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include 45 Hashimoto's patients attending the out clinics of Endocrinology Department of Assiut university hospital. In addition, 45 healthy blood donors will be included as controls. The diagnosis of hashimoto's thyroiditis will be determined according to the criteria of American Thyroid Association;
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Measure the frequency of Follicular helper Tcells and Follicular regulatory T cells in peripheral blood samples in Hashimoto's pts in comparison with control. | Baseline
  Measure changes in number of surface markers CD4 , ICOS, CXCR5 and FOXP3. Follicular helper Tcells and Follicular regulatory T cells in peripheral blood samples in Hashimoto's pts in comparison with control.

REFERENCES:
- See also: Mincer DL, Jialal I. Hashimoto Thyroiditis. [Updated 2023 Jul 29]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2024 Jan- — http://www.ncbi.nlm.nih.gov/books/NBK459262/